CLINICAL TRIAL: NCT01845168
Title: Prevention of Peptic Ulcer Bleeding Related to the Use of NSAIDs and Aspirin by Using "Computer-alert" - a Randomized Study in General Practice
Brief Title: Prevention of Gastric Ulcer Bleeding by Using "Computer-alert" in General Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Johanna Petersen, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20120034
Record Dates: First submitted 2013-03-13; First posted 2013-05-03 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Bleeding Peptic Ulcer
Keywords: Bleeding peptic ulcer; NSAID and Aspirin; Computer-alert; General practitioner
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer-alert (Active Comparator): 2 arm study active group: 'A computer alert which pops up when the GP prescribes NSAID/ASA to a patient with risk-factors
  Interventions: Other: Computer-alert; Device: A computer alerts which pops up when the GP presribes NSAID/ASA to a patient with risk-factors; Device: Computer-alert
- controlgroup, normal procedures (No Intervention): The control-group: GP working in normal procedures

INTERVENTIONS:
Other: Computer-alert — A computer-alert which is activated when the physician is making a prescription for ASA or NSAID. Only for patients with riskfactors such as: Age over 60, males-gender, NSAID and ASA in kombination, Adenosine-diphosphate-inhibitor (ADP-inhibitor), blood-thinning medicine, Selective serotonin reuptake-inhibitor (SSRI) and steroids
  Arms: Computer-alert
Device: A computer alerts which pops up when the GP presribes NSAID/ASA to a patient with risk-factors — A computer-alert which is activated when the physician is making a prescription for ASA or NSAID. Only for patients with riskfactors such as: Age over 60, males-gender, NSAID and ASA in combination, ADP-inhibitor, bloodthinning medicine, SSRI, and steroids
  Arms: Computer-alert
Device: Computer-alert
  Arms: Computer-alert

SUMMARY:
The purpose of this study is to investigate if a computerised decision-support tool used in general practice, can reduce the frequency of peptic ulcer bleeding related to the use of NSAIDs (Non-Steroidal-antiinflammatory-drug) and ASA( Acetylsalicylic acid) .

On the basis of "The Danish general medical database" it is possible to develope a computerised decision-support tool, which enables the general practitioner (GP) in a "pop-up" window to get information on each patients risk-factors, when prescribing NSAID and aspirin to a patient at risk. This will give the general practitioner the oppurtunity to choose a different type of preparation or prescribe ulcer-preventive medicine at the same time.

The decision-support tool will be tested in a randomized trial among general practitioners. The aim is to reduce the occurence of peptic ulcer bleeding. The expected outcome is a reduction in half of the total numbers of peptic ulcers.

DETAILED DESCRIPTION:
The background of the study is that NSAIDs and Aspirins increase the risk of peptic ulcer bleeding. On average 1-2% of patients using NSAID and Aspirin will develope gastric ulcer bleeding. But for patients with one or more risk-factors, the risk increases to 9% per 6 months. The mortality in this case is 10-15%. Approximately 3200 patients are admitted to the hospital with bleeding ulcer annually in Denmark.

Danish investigations have shown that 80% of all peptic ulcer bleedings admitted to hospital are related to the use of NSAID or Aspirin.

The consumption of NSAID and Aspirin is large. A third of people over 60 are treated within a year with these preparations. The risk of developing gastric ulcer related to NSAID and Aspirin can be reduced by concomitant therapy with antacids. Several studies have shown that only 20-30% of patients with risk-factors receive ulcer preventive medicine.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners in the Region of Southern Denmark which are linked to Danish General Medical Database for minimum 6 months

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-02 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Patient outcome: The number of hospitalizations due to bleeding ulcer complication. | one year

SECONDARY OUTCOMES:
Patient outcome: The number of uncomplicated ulcer diagnosed by endoscopy. | one year

OTHER OUTCOMES:
Prescription changes: How often the GP refrains the ASA/NSAID-treatment because of the risk-information and the computer-alert | one year
Prescription changes: The number of patients with riskfactors, who will recieve a prescription of ulcer preventive medicine | one year
Prescription changes: general changes in the frequency of NSAID ordinations | one year

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Petersen, MD, Principal Investigator — Afdeling for medicinske mavetarmsygdomme, Odense Universitetshospital.; Jane M Hansen, MD, Ph.D, Study Director — Afdeling for Medicinske mavetarmsygdomme; Johanna M Petersen, MD, Principal Investigator — Afdeling for medicinske mavetarmsygdomme, Odense Universitetshospital
Locations (2):
- Denmark (2):
  - Afdeling for medicinske mavetarmsygdomme - Odense Universitetshospital, Odense, Funen
  - Afdeling for medicinske mavetarmsygdomme, Odense Universitetshospital, Odense